CLINICAL TRIAL: NCT04841928
Title: Optimization of Psychological Treatment for Pain After Breast Cancer Using the Multiphase Optimization Strategy (MOST): A Pilot Study
Brief Title: Optimizing Psychological Treatment for Pain After Breast Cancer: A Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Danish Council for Independent Research (Other)
Responsible Party: Principal Investigator, Maja Johannsen, Assistant Professor, University of Aarhus
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: MOST Pain Pilot
Record Dates: First submitted 2021-03-23; First posted 2021-04-12 (Actual); Last update posted 2021-09-30 (Actual); Status verified 2021-09

CONDITIONS: Pain, Chronic; Breast Cancer
Keywords: Breast cancer; Pain; Third wave cognitive therapy; Mindful attention; Decentering; Values and committed action; The Multiphase Optimization Strategy (MOST); Psychological pain treatment; Treatment mediators
MeSH Terms: conditions — Chronic Pain; Breast Neoplasms; Pain

STUDY DESIGN:
Intervention Model Description: The study uses a 2^3 factorial design, randomizing participants to 8 experimental conditions
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (8):
- Waitlist control (No Intervention): Participants randomized to condition 1 are not offered any treatment components immediately upon enrollment, but will be offered a treatment component of own choice at the end of the study. Total number of sessions: 2 (2 contact hours) following study completion.
- Mindful attention (Experimental): Participants randomized to condition 2 will receive the Mindful attention treatment component. Total number of sessions: 2 (2 contact hours).
  Interventions: Behavioral: Mindful attention
- Decentering (Experimental): Participants randomized to condition 3 will receive the Decentering treatment component. Total number of sessions: 2 (2 contact hours).
  Interventions: Behavioral: Decentering
- Values and committed action (Experimental): Participants randomized to condition 4 will receive the Values and committed action treatment component. Total number of sessions: 2 (2 contact hours).
  Interventions: Behavioral: Value-based action
- Mindful attention + Decentering (Experimental): Participants randomized to condition 5 will receive the Mindful attention treatment component and the Decentering treatment component. Total number of sessions: 4 (4 contact hours).
  Interventions: Behavioral: Mindful attention; Behavioral: Decentering
- Mindful attention + Values and committed action (Experimental): Participants randomized to condition 6 will receive the Mindful attention treatment component and the Values and committed action treatment component. Total number of sessions: 4 (4 contact hours).
  Interventions: Behavioral: Mindful attention; Behavioral: Value-based action
- Decentering + Values and committed action (Experimental): Participants randomized to condition 7 will receive the Decentering treatment component and the Values and committed action treatment component. Total number of sessions: 4 (4 contact hours).
  Interventions: Behavioral: Decentering; Behavioral: Value-based action
- Mindful attention + Decentering + Value-based action (Experimental): Participants randomized to condition 8 will receive the Mindful attention treatment component, the Decentering treatment component, and the Values and committed action treatment component. Total number of sessions: 6 (6 contact hours).
  Interventions: Behavioral: Mindful attention; Behavioral: Decentering; Behavioral: Value-based action

INTERVENTIONS:
Behavioral: Mindful attention — The Mindful attention treatment component consists of a breathing exercise and is operationalized as two sessions (1 hour each) delivered over two weeks, i.e., one session per week, with homework between sessions. Sessions will be delivered online.
  Arms: Mindful attention; Mindful attention + Decentering; Mindful attention + Decentering + Value-based action; Mindful attention + Values and committed action
Behavioral: Decentering — The Decentering treatment component consists of a guided imagery exercise and is operationalized as two sessions (1 hour each) delivered over two weeks, i.e., one session per week, with homework between sessions. Sessions will be delivered online.
  Arms: Decentering; Decentering + Values and committed action; Mindful attention + Decentering; Mindful attention + Decentering + Value-based action
Behavioral: Value-based action — The Values and committed action treatment component consists of identification of personal values and committed action, and is operationalized as two sessions (1 hour each) delivered over two weeks, i.e., one session per week, with homework between sessions. Sessions will be delivered online.
  Arms: Decentering + Values and committed action; Mindful attention + Decentering + Value-based action; Mindful attention + Values and committed action; Values and committed action

SUMMARY:
The present study is a pilot study that aims to evaluate the feasibility, validity, and preliminary efficacy of three psychological treatment components for pain after breast cancer, which will be evaluated in a larger trial following completion of the present pilot study.

DETAILED DESCRIPTION:
The present pilot study is a precursor for a following larger trial and aims to evaluate the i) feasibility, ii) validity, and iii) preliminary efficacy of the three treatment components that will be further investigated in a subsequent larger trial. The present pilot study will employ the same design as will be used in the subsequent larger trial, namely the Multiphase Optimization Strategy (MOST). Specifically, in the subsequent larger trial, MOST will be used to evaluate the efficacy and change processes of three psychological treatment components selected from so-called "third wave" cognitive therapies (CTs), which have been shown to be efficacious in the treatment of pain after breast cancer.

The overall hypothesis is that the selected third wave CT components will target key maintaining psychological factors in pain, thus leading to reductions in the primary outcomes of pain intensity and -interference. Specifically, we hypothesize that:

1. Mindful attention practices will increase attentional control (i.e., the ability to intentionally focus and intentionally shift one's attention), thereby reducing pain hypervigilance, leading to reductions in pain intensity and -interference.
2. Decentering practices will reduce fusion with thoughts (i.e., getting caught up in one's thoughts and acting automatically in response to thoughts), thereby reducing pain catastrophizing, leading to reductions in pain intensity and -interference.
3. Values and committed action (i.e., behavior linked to values and goals) will increase acceptance of discomfort and reduce avoidant behavior, leading to reductions in pain intensity and -interference.

ELIGIBILITY:
Inclusion criteria:

* Diagnosis of primary breast cancer stage I-III
* Min. 6 months post breast cancer treatment (i.e., surgery, chemotherapy, and/or radiotherapy). Endocrine treatment, e.g., Letrozole or Tamoxifen, and/or Zoledronic acid and/or Herceptin treatment is allowed during study participation
* Pain corresponding to a min. pain score of >= 3 on pain intensity or pain interference measured by 11-point Numeric Rating Scales (NRSs)
* Sufficient ability to communicate in Danish
* Sufficient ability to participate in an online-delivered intervention

Exclusion Criteria:

* Metastatic breast cancer (stage IV)
* Breast cancer recurrence
* Bilateral breast cancer
* Other current cancer disease
* Other current pain condition (e.g., fibromyalgia)
* Current severe psychiatric disorder (e.g., psychosis)
* Inability to communicate in Danish
* Inability to participate in an online-delivered intervention

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
Pain intensity (11-point Numeric Rating Scale, NRS) | Baseline (T1) to 1 week after last session (Post-intervention, T2)
  The NRS is a validated, self-report instrument assessing pain intensity during the last week. Answer format range: 0 (no pain) to 10 (worst possible pain); total score range: 0-10. Higher scores yield more pain.
Pain interference (the 7-item subscale of the Brief Pain Inventory, BPI) | Baseline (T1) to 1 week after last session (Post-intervention, T2)
  The BPI is a validated, self-report instrument assessing clinical pain. The BPI pain interference subscale assesses pain interference during the last week across 7 domains, i.e., general activity, mood, walking ability, normal work, relations with other people, sleep, and enjoyment of life. Answer format range: 0 (no interference) to 10 (maximal interference); total score range: 0-10. Higher scores yield more pain interference.

SECONDARY OUTCOMES:
Pain intensity (11-point Numeric Rating Scale, NRS) | Every day for 6 days following the first session (Td) for each treatment component
  Pain intensity during the last 24 hours will be assessed every day for 6 days following the first session (Td) for each treatment component using the NRS. Answer format range: 0 (no pain) to 10 (worst possible pain); total score range: 0-10. Higher scores yield more pain.
4. Pain interference (1 aggregated item assessing pain interference during the last 24 hours within the 7 domains measured with the Brief Pain Inventory, BPI, interference subscale) | Every day for 6 days following the first session (Td) for each treatment component
  Pain interference during the last 24 hours will be assessed every day for 6 days following the first session (Td) for each treatment component using 1 aggregated item assessing pain interference across the 7 domains measured with the BPI interference subscale, i.e., general activity, mood, walking ability, normal work, relations with other people, sleep, and enjoyment of life. Answer format range: 0 (no interference) to 10 (maximal interference); total score range: 0-10. Higher scores yield more pain interference.
Pain burden (11-point Numeric Rating Scale, NRS) | Baseline (T1) to 1 week after last session (Post-intervention, T2)
  The NRS is a validated, self-report instrument assessing pain burden during the last week. Answer format range: 0 (no burden) to 10 (maximal burden); total score range: 0-10. Higher scores yield more pain burden.
Pain quality (the 22-item pain descriptors from the McGill Pain Questionnaire, MPQ) | Baseline (T1) to 1 week after last session (Post-intervention, T2)
  The pain descriptors from the MPQ constitutes a validated, self-report instrument assessing pain quality (i.e., pain type, namely continuous pain, intermittent pain, neuropathic pain, affective pain) during the last week. Answer format range: 0 (no pain) to 10 (worst possible pain); total score range: 0-60 (continuous, neuropathic and intermittent pain), 0-40 (affective pain). Higher scores yield more pain.
Pain catastrophizing (the 13-item Pain Catastrophizing Scale, PCS) | Baseline (T1) to 1 week after last session (Post-intervention, T2)
  The PCS is a validated, self-report instrument assessing pain catastrophizing. Answer format range: 0 (not at all) to 4 (all the time); total score range: 0-52. Higher scores yield more pain catastrophizing.
Psychological distress (the 14-item Hospital Anxiety and Depression Scale, HADS) | Baseline (T1) to 1 week after last session (Post-intervention, T2)
  The HADS is a validated, self-report instrument assessing psychological distress during the last week. Answer format range: 0 (not at all or never) to 3 (most or all of the time); total score range 0-42. Higher scores yield more distress.
Fear of cancer recurrence (the 9-item Fear of Cancer Recurrence Inventory, FCRI) | Baseline (T1) to 1 week after last session (Post-intervention, T2)
  The FCRI is a validated, self-report instrument assessing fear of cancer recurrence during the last month. Answer format range: 0 (not at all) to 4 (a great deal); total score range 0-36. Higher scores yield more fear of cancer recurrence.
Well-being (the 5-item WHO-5 Well-Being Index, WHO-5) | Baseline (T1) to 1 week after last session (Post-intervention, T2)
  The WHO-5 is a validated, self-report instrument assessing current well-being. Answer format range: 0 (at no time) to 5 (all the time); total score range: 0-100. Higher scores yield more well-being.

OTHER OUTCOMES:
Qualitative Interviews | 10-14 days after last session
  Participants will be invited to participate in a 30-minutes semi-structured individual interview 10-14 days after their last session. The interview serves to support the validation of the treatment components and to provide in-depth knowledge about the participants' experiences through their qualitative comments.
Moderator: Demographic characteristics | Baseline (T1)
  Socio-demographic characteristics will be assessed using single questions (e.g., municipality, marital status, income, work status).
Moderator: Clinical characteristics | Baseline (T1)
  Clinical characteristics will be assessed using single questions (e.g., date of surgery, adjuvant therapy).
Moderator: Treatment expectancy | Baseline (T1)
  Treatment expectancy will be assessed using a single question regarding the extent to which the participant believes that the intervention will reduce pain and increase overall well-being. Answer format range: 1 (not at all) to 5 (a great deal); total score range: 1-5. Higher scores indicate stronger expectations that the intervention will lead to a positive outcome.
Moderator: Therapeutic alliance (the 12-item Working Alliance Inventory, WAI) Revised Short Form | 1 week after last session (Post-intervention, T2)
  The WAI is a validated, self-report instrument assessing therapeutic alliance. Answer format range: 1 (never) to 7 (all the time); total score range: 12-84. Higher scores yield a stronger therapeutic alliance.
Moderator: Home work | Before each session (Ts) and 1 week after last session (Post-intervention, T2)
  Homework will be assessed with 4 single items related to i) whether home work has been conducted (yes/no), and the ii) type, iii) frequency (number of days per week), and iv) duration of completed homework (average number of minutes per day).
Mediator: Mindful attention (the 15-item Mindful Attention Awareness Scale, MAAS) | Baseline (T1) to 1 week after last session (Post-intervention, T2)
  The MAAS is a validated, self-report instrument assessing individual differences in the frequency of mindful states over time. Answer format range: 1 (almost always) to 6 (almost never); total score range: 1-6. Higher scores yield higher levels of mindful attention.
Mediator: Mindful attention (2 items from the 15-item Mindful Attention Awareness Scale, MAAS) | Before each session (Ts)
  MAAS items 13 and 7 will be assessed before each session (Ts). Answer format range: 1 (almost always) to 6 (almost never). Higher scores yield higher levels of mindful attention.
Mediator: Mindful attention (1 item from the 15-item Mindful Attention Awareness Scale, MAAS) | Every day for 6 days following the first session for each treatment component (Td)
  MAAS item 6 will be assessed every day for 6 days following the first session (Td) for each treatment component. Answer format range: 1 (almost always) to 6 (almost never). Higher scores yield higher levels of mindful attention.
Mediator: Decentering (the 11-item subscale of the Experiences Questionnaire, EQ) | Baseline (T1) to 1 week after last session (Post-intervention, T2)
  The EQ is a validated, self-report instrument assessing decentering. Answer format range: 1 (do not agree at all) to 5 (agree completely); total score range: 11-55. Higher scores yield higher levels of decentering.
Mediator: Decentering (2 items from the 11-item subscale of the Experiences Questionnaire, EQ) | Before each session (Ts)
  EQ items 5 and 7 will be assessed before each session (Ts). Answer format range: 1 (do not agree at all) to 5 (agree completely). Higher scores yield higher levels of decentering.
Mediator: Decentering (1 item from the 11-item subscale of the Experiences Questionnaire, EQ) | Every day for 6 days following the first session for each treatment component (Td)
  EQ item 5 will be assessed every day for 6 days following the first session (Td) for each treatment component. Answer format range: 1 (do not agree at all) to 5 (agree completely). Higher scores yield higher levels of decentering.
Mediator: Pain acceptance and activity engagement (the 20-item Chronic Pain Acceptance Scale, CPAS) | Baseline (T1) to 1 week after last session (Post-intervention, T2)
  The CPAS is a validated, self-report instrument assessing pain acceptance and activity engagement. Answer format range: 0 (never true) to 6 (always true); subscale score range: 0-54 (pain acceptance subscale), 0-66 (activity engagement subscale). Higher scores yield more acceptance and activity engagement.
Mediator: Pain acceptance and activity engagement (2 items from the 20-item Chronic Pain Acceptance Scale, CPAS) | Before each session (Ts)
  CPAS items 1 and 12 will be assessed before each session (Ts). Answer format range: 0 (never true) to 6 (always true). Higher scores yield more acceptance and activity engagement.
Mediator: Pain acceptance and activity engagement (1 item from the 20-item Chronic Pain Acceptance Scale, CPAS) | Every day for 6 days following the first session for each treatment component (Td)
  CPAS item 1 will be assessed every day for 6 days following the first session (Td) for each treatment component. Answer format range: 0 (never true) to 6 (always true). Higher scores yield more acceptance and activity engagement.

CONTACTS AND LOCATIONS:
Overall Officials: Maja Johannsen, PhD, Principal Investigator — University of Aarhus
Locations (1):
- Aarhus University, Aarhus, Central Jutland, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Buskbjerg CR, Johannsen M, Norskov CC, Jensen AB, Frederiksen Y, Egerod I, Guastaferro K, Johansen C, von Heymann A, Speckens A, O'Toole MS, Zachariae R. Optimizing Psychological Treatment for Pain After Breast Cancer Using a Randomized Factorial Design: A Feasibility Study. Scand J Psychol. 2025 Dec 31. doi: 10.1111/sjop.70063. Online ahead of print. PMID 41474052